CLINICAL TRIAL: NCT05422638
Title: Fostering Resilience to Race-Based Stress: A Pilot Study
Brief Title: Race-Based Stress Trauma and Empowerment
Acronym: RBSTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D4070-P; 1I21RX004070-01A1 (NIH)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Life Stress; Racism
Keywords: Life stress; Racism; Health promotion; Randomized controlled trial
MeSH Terms: conditions — Stress, Psychological; Racism

STUDY DESIGN:
Intervention Model Description: RBSTE is a group-based approach that combines cultural adaptations of established psychotherapeutic techniques with novel strategies to foster resilience and empowerment for VOC.
  PCT is a group-based approach that provides a safe space for VOC to discuss stressors and find adaptive of responding to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RBSTE (Experimental): 8-week health promotion group focused on supporting coping with racism and empowerment
  Interventions: Behavioral: RBSTE
- PCT (Active Comparator): 8-week health promotion group focused on providing support and facilitating problem solving
  Interventions: Behavioral: PCT

INTERVENTIONS:
Behavioral: RBSTE — 8-week health promotion group focused on supporting coping with racism and empowerment
  Arms: RBSTE
Behavioral: PCT — 8-week health promotion group focused on providing support and facilitating problem solving
  Other Names: Present Centered Therapy
  Arms: PCT

SUMMARY:
The existence of racially/ethnically based health disparities is well established, both within the civilian community and among Service Members and Veterans. Experiences of discrimination are acute and chronic stressors that substantially contribute to greater emotional distress, poorer health behavior, lower healthcare utilization and increased allostatic load, all of which undermine well-being, functioning and Whole Health. An innovative clinical program, the Race-Based Stress/Trauma and Empowerment (RBSTE) group, was developed to help Veterans of Color to build coping resources and empowerment. Although qualitative data suggest the promise of this intervention, systematic evaluation is lacking. The proposed feasibility project will lay the groundwork for a future randomized controlled trial to evaluate RBSTE as compared to a control group in terms of Whole Health, functioning and mental/physical wellness. The project thus begins a program of research to address the health implications of systemic racism.

DETAILED DESCRIPTION:
Health disparities between White and Black, Indigenous and People of Color (BIPOC) are well documented in the United States; this phenomenon is driven in part by discrimination experiences and is an important contributor to well-being and functioning, including among military service members and Veterans. The chronic stress of racism has both psychological and physiological effects. Discrimination is associated with increased psychological distress, including higher rates of PTSD among Veterans of Color (VOC), poorer health behavior and decreased healthcare utilization. Race-based stress is also linked to increased allostatic load (AL), which is a measurable index of wear-and-tear on the body due to chronic stress exposure that is associated with greater disease burden and mortality. Recognizing the unmet need for interventions to help VOC process and cope with experiences of discrimination, the Race-based Stress/Trauma and Empowerment (RBSTE) intervention (Carlson, Endsley, Motley, Shawahin, & Williams, 2018) was developed. RBSTE is a group-based approach that combines cultural adaptations of established psychotherapeutic techniques with novel strategies to foster resilience and empowerment for VOC. Initial qualitative data suggests the promise of this approach, but no systematic data are yet available to determine whether or not RBSTE is achieving its goals of enhancing coping and restoring well-being. The proposed project is a pilot randomized controlled trial (RCT) with multi-modal longitudinal assessment. Participants will be recruited from VA facilities and the surrounding community. VOC who report race-based stress, with minimal exclusions, will be evaluated at baseline, randomized in groups to one of two wellness interventions and then re-evaluated immediately after treatment. The interventions include RBSTE and Present Centered Therapy (PCT), designed to control for nonspecific aspects of RBSTE, including support and participation in an all-BIPOC group. The interventions will be delivered in 8 weekly 90-minute group sessions by a trained mental health professional using videoconferencing. The aims of the project are (1) to assess the feasibility of recruiting VOC for an RCT of this nature; (2) to examine the acceptability and appropriateness of intervention content, the feasibility of participation, and participant's perceptions of provider behavior and attitudes; and (3) to establish the optimal strategy for quantifying mental and physical health outcomes for future studies. Thus, the project will set the stage for evaluation of RBSTE's efficacy and ultimately implementation. This critically important program of research will provide guidance as to best practices for the management of race-based stress, with the ultimate goal of eliminating health disparities for Veterans and the community more broadly.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as a BIPOC
* Veteran
* able to consent to study activities
* endorsing one or more perceived discrimination experiences on the Everyday Discrimination Form (short version) or the Major Experiences of Discrimination Scale (abbreviated version) "a few times a year" or more frequently and endorsing stress on a validated single-item measure

Exclusion Criteria:

* serious mental illness, alcohol/substance use disorders, or cognitive impairment that may interfere with the ability to benefit from group

  * (e.g., severe depression, psychotic illness, mania, dementia, untreated alcohol/substance dependence)
* serious suicidality or homicidality (e.g., ideation with plan/intent) that is likely to require urgent/emergent intervention within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J. Lang, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Malaktaris A, McLean CL, Kelsven S, Chu GM, Ross KS, Endsley M Jr, Minassian A, Liu L, Hong S, Lang AJ. Mitigating the health effects of systemic racism: Evaluation of the Race-Based Stress and Trauma Empowerment intervention. Contemp Clin Trials. 2023 Apr;127:107118. doi: 10.1016/j.cct.2023.107118. Epub 2023 Feb 14. PMID 36796623

RESULTS

PARTICIPANT FLOW:
Groups:
- Race-Based Stress Trauma & Empowerment (RBSTE): 8-week health promotion group focused on supporting coping with racism and empowerment
  RBSTE: 8-week health promotion group focused on supporting coping with racism and empowerment
- Present-Centered Wellness Group (PCWG): 8-week health promotion group focused on providing support and facilitating problem solving
  PCWG: 8-week health promotion group focused on providing support and facilitating problem solving
Period: Overall Study
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Started | 19 | 18
Completed (Completion of at least 5 intervention sessions) | 11 | 16
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- PCWG: 8-week health promotion group focused on providing support and facilitating problem solving
  PCWG: 8-week health promotion group focused on providing support and facilitating problem solving
- Total: Total of all reporting groups
Arm/Group | RBSTE | PCWG | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (17) | 46.9 (14.6) | 49.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 4 | 5 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Percentage of individuals enrolled out of total contacted
Time Frame: week 0
Measure: Number; unit: percentage of individuals approached
Groups:
- Total Sample: All individuals approached about the study
Arm/Group | Total Sample
Number analyzed (Participants) | 417
percentage of individuals approached | 8.87

2. Primary Outcome: Initiation Rate
Description: Percentage of subjects who initiate any intervention among all enrolled subjects
Time Frame: week 1
Population: Participants did not know their condition until they arrived for the first session, so these data should not be interpreted by group.
Measure: Number; unit: percentage of enrolled individuals
Groups:
- RBSTE: Individuals who enrolled for the study and were assigned to RBSTE
- PCWG: Individuals who were enrolled in the study and assigned to PCWG
Arm/Group | RBSTE | PCWG
Number analyzed (Participants) | 19 | 18
percentage of enrolled individuals | 73.7 | 100

3. Primary Outcome: Per Protocol Completion
Description: Percentage of subjects who complete 5 or 6 sessions of intervention among those who start the intervention
Time Frame: week 8
Population: Includes the 34 participants of the 37 enrolled who initiated intervention.
Measure: Number; unit: percent inititiators completed 5+
Arm/Group | RBSTE | PCWG
Number analyzed (Participants) | 17 | 17
percent inititiators completed 5+ | 64.7 | 94.1

4. Primary Outcome: Intent-to-treat Completion
Description: Percentage of subjects who complete 5 or 6 sessions of intervention among all randomized subjects
Time Frame: week 8
Measure: Number; unit: percentage of ITT completed 5+
Arm/Group | RBSTE | PCWG
Number analyzed (Participants) | 19 | 18
percentage of ITT completed 5+ | 57.9 | 88.9

5. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Perceived acceptability of the interventions by participants AIM range 4-20 with greater scores indicating better acceptability
Time Frame: week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 7 | 8
total score on a scale | 18.43 (1.81) | 14.75 (3.84)

6. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: Perceived appropriateness of the interventions by participants IAM range 4-20 with greater scores indicating better appropriateness
Time Frame: week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 7 | 8
total score on a scale | 17.57 (2.70) | 14.25 (3.77)

7. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: Perceived feasibility of the interventions by participants FIM range 4-20 with greater scores indicating better feasibility
Time Frame: week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 7 | 8
total score on a scale | 17.43 (2.22) | 14.88 (3.52)

8. Secondary Outcome: Brief Personal Health Inventory (B-PHI): Physical Health
Description: self-appraisal of physical well being range 1-5 with higher scores indicating better health
Time Frame: change from week 1 to week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 10 | 8
change score on a scale | 0.1 (0.88) | 0.27 (0.53)

9. Secondary Outcome: Brief Personal Health Inventory (B-PHI): Mental Health
Description: self-appraisal of mental well being range 1-5 with higher scores indicating better mental health
Time Frame: change from week 1 to week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 10 | 8
change in score on a scale | 0.97 (1.14) | 0.61 (0.76)

10. Secondary Outcome: Brief Personal Health Inventory (B-PHI): Daily Living
Description: self-appraisal of daily living range 1-5 with higher scores indicating better daily living
Time Frame: change from week 1 to week 8
Population: Reduced numbers reflect missing data
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
Number analyzed (Participants) | 10 | 8
change in score on a scale | 1.07 (0.99) | 0.43 (0.93)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Race-Based Stress Trauma & Empowerment (RBSTE) | Present-Centered Wellness Group (PCWG)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT05422638/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT05422638/ICF_000.pdf